CLINICAL TRIAL: NCT04498767
Title: Stereotactic Body Radiotherapy in Addition to Standard of Care Treatment in Patients With Rare Oligometastatic Cancers (OligoRARE): a Randomized, Phase 3, Open-label Trial
Brief Title: Stereotactic Body Radiotherapy in Patients With Rare Oligometastatic Cancers (OligoRARE)
Acronym: OligoRARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Anticancer Fund, Belgium (Other); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 1945
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Gynecologic Cancer; Skin Cancer; Head and Neck Cancer; Sarcoma; Renal Cancer; Bladder Cancer; Upper Urinary Tract Carcinoma; Pancreatic Cancer; Hepatobiliary Cancer; Gastric Cancer; Small Bowel Cancer; Esophageal Cancer; Melanoma; Colon Cancer; Oligometastasis
Keywords: oligometastatic cancer; Stereotactic body radiotherapy; SBRT
MeSH Terms: conditions — Skin Neoplasms; Head and Neck Neoplasms; Sarcoma; Kidney Neoplasms; Urinary Bladder Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Melanoma; Colonic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Standard of Care + palliative RT (Active Comparator): Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications. Recommended dose fractionations in this arm will include 8 Gy in 1 fractions, 20 Gy in 5 fractions, and 30 Gy in 10 fractions. Patients in this arm should not receive stereotactic doses or radiotherapy boosts, unless there is a clearly known clinical benefit (e.g. stereotactic radiation to a new brain metastases when all disease is controlled on systemic therapy).
  Systemic therapy will be pre-specified based on the standard of care approach for that patient, and it may include cytotoxic, targeted, hormonal, or immunotherapy.
  Interventions: Radiation: Palliative RT
- Arm 2: Standard of Care + SBRT (Experimental): The experimental arm consists of SBRT (and standard of care systemic therapy). Each lesion may be treated with 1, 3, or 5 SBRT fractions of 16-24 Gy, 24-33 Gy or 25-40 Gy, respectively, depending on the local practice and size & location of oligometastases. Three-fraction regimens will deliver a fraction every second day, and five-fraction regimens are delivered daily. All treatments must be completed within 2 weeks (10 working days) in order to avoid delays in starting systemic therapy.
  Patients treated with prior or concomitant systemic therapy are eligible for this study. Use of chemotherapy regimens, targeted therapy or immunotherapy containing potent enhancers of radiation damage (e.g. gemcitabine, doxorubicin) can be postponed or interrupted for a duration of one month after radiation.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Each lesion may be treated with 1, 3, or 5 SBRT fractions of 16-24 Gy, 24-33 Gy or 25-40 Gy, respectively, depending on the local practice and size & location of oligometastases. Three-fraction regimens will deliver a fraction every second day, and five-fraction regimens are delivered daily. All treatments must be completed within 2 weeks (10 working days) in order to avoid delays in starting systemic therapy.
  Other Names: SBRT
  Arms: Arm 2: Standard of Care + SBRT
Radiation: Palliative RT — Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications. Recommended dose fractionations in this arm will include 8 Gy in 1 fractions, 20 Gy in 5 fractions, and 30 Gy in 10 fractions. Patients in this arm should not receive stereotactic doses or radiotherapy boosts, unless there is a clearly known clinical benefit (e.g. stereotactic radiation to a new brain metastases when all disease is controlled on systemic therapy).
  Arms: Arm 1: Standard of Care + palliative RT

SUMMARY:
This is a randomized open-label multicentre Phase III superiority study of the effect of adding SBRT to the standard of care treatment on overall survival in patients with rare oligometastatic cancers.

Patients will be randomized in a 1:1 ratio between current standard of care treatment vs. standard of care treatment + SBRT to all sites of known metastatic disease.

The primary objective of this trial is to assess if the addition of stereotactic body radiotherapy (SBRT) to standard of care treatment improves overall survival (OS) as compared to standard of care treatment alone in patients with rare oligometastatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* Controlled primary tumour, defined as:
* at least 3 months since original tumour treated definitively, with no progression at primary site
* Total number of oligometastases of 1-5 including:
* Brain metastases amenable to radiosurgery or fractionated stereotactic radiotherapy patient who had neurosurgical resection before trial inclusion are allowed and resected brain metastases count to the total number of oligometastases
* All sites of disease can be safely treated based on the judgement of an experienced radiation oncologist
* ECOG score 0-2
* Life expectancy > 6 months
* Age 18 or older
* Before patient randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Primary cancer of prostate, breast, lung or colorectal
* Serious medical comorbidities precluding radiotherapy:
* These include interstitial lung disease in patients requiring thoracic radiation, Crohn's disease in patients where the GI tract will receive radiotherapy, or ulcerative colitis where the bowel will receive radiotherapy and connective tissue disorders such as lupus or scleroderma.
* For patients with liver metastases, moderate/severe liver dysfunction (Child Pugh B or C)
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated previously with radiation, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed in the RTQA Guidelines. All such cases should be discussed with one of the study coordinators
* Brain metastases only, without extra-cerebral metastases
* Malignant pleural effusion, malignant ascites, meningeal carcinomatosis and peritoneal carcinomatosis
* Maximum size of 6 cm for lesions outside the brain, except:
* Bone metastases over 5 cm may be included, if in the opinion of the local radiation oncologist it can be treated safely (e.g. rib, scapula, pelvis)
* Clinical or radiologic evidence of symptomatic spinal cord compression. Patients can be eligible if surgical resection has been performed, but the surgical site counts toward the total of up to 3 metastases.
* Metastatic disease that invades any of the following: GI tract (including oesophagus, stomach, small or large bowel), mesenteric lymph nodes, or disseminated skin metastases and lymphangiosis
* Pregnant or breast feeding women
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 7.5 years from first patient in
  Overall survival is the time interval from the date of randomization to the date of death whatever the cause of death. Patients who are alive are censored at the last date known to be alive.

SECONDARY OUTCOMES:
Progression-free survival | 9 years from first patient in
Disease-specific survival | 9 years from first patient in
Time to disease progression | 9 years from first patient in
  Disease-specific survival is the time interval from the date of randomization to the date of cancer-related death.
Time to development of new metastatic lesions | 9 years from first patient in
  Time to development of new metastatic lesions is the time interval from the date of randomization to the date of first occurrence of any of the following events:
  * Development new metastatic lesions,
  * Cancer-related death.
Time to development of polymetastatic disease | 9 years from first patient in
  Time to development of polymetastatic disease is the time interval from the date of randomization to the date of first occurrence of any of the following events:
  * Presence of more than 5 metastases at a specific timepoint during follow-up,
  * Development of metastases that preclude treatment with SBRT (e.g. due to large size or locating in previously irradiated region where re-irradiation is not possible),
  * Cancer-related death.
Adverse events graded according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0 | 9 years from first patient in
Health-related quality of life evaluated using self-administered EORTC QLQ-C30 questionnaires | 9 years from first patient in
Health-related quality of life evaluated using self-administered EQ-5D-5L questionnaires | 9 years from first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Principal Investigator — University of Zurich; Piet Ost, Principal Investigator — Gasthuiszusters Antwerpen - Sint-Augustinus
Locations (13):
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Gent, Ghent
  - Gasthuiszusters Antwerpen - Sint-Augustinus, Wilrijk
- France (2):
  - Centre Oscar Lambret, Lille
  - Gustave Roussy, Villejuif
- Universitaets Krankenhaus Eppendorf - Universitaetsklinikum Hamburg-Eppendorf KE - University Cancer Center, Hamburg, Martinistrasse 52, Germany
- Istituto Europeo di Oncologia, Milan, Italy
- Poland (2):
  - Medical University Of Gdansk, Gdansk, Mariana Smoluchowskiego 17
  - Maria Sklodowska-Curie Memorial Cancer Centre - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Switzerland (2):
  - Inselspital, Bern
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust (UHB) - UHB-Queen Elisabeth Medical Centre, Birmingham
  - Royal Marsden Hospital - site: Chelsea, London, London